CLINICAL TRIAL: NCT07309926
Title: Comparative Analysis of Spatiotemporal Gait Parameters and Paraspinal Surface Electromyography Parameters in Degenerative Spinal Diseases: A Cross-Sectional Study Using Motion Capture and Electromyographic Ensemble Averaging
Brief Title: Gait and Paraspinal sEMG in Degenerative Spinal Diseases
Acronym: TDGKSEPDSD
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: xuanwu_DSD
Record Dates: First submitted 2025-05-20; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-05

CONDITIONS: Adult Spinal Deformity; Degenerative Scoliosis; Sagittal Deformity; Sagittal Imbalance; Coronal Vertical Axis; Lumbar Spinal Stenosis; Lumbar Disc Herniation; Cervical Spondylosis With Myelopathy
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Degenerative Scoliosis Group: This group comprised elderly patients (>60 years old) diagnosed with degenerative lumbar scoliosis (DLS) (Cobb angle >20°). Patients were excluded if they had concurrent neurological disorders, other spinal pathologies, or lower limb conditions that could influence gait mechanics. Additionally, individuals with a history of spinal or lower limb surgery were also excluded to minimize confounding factors.
  Interventions: Other: Gait analysis and surface electromyography analysis
- Sagittal Imbalance Group: This group comprised elderly patients (>60 years old) diagnosed with sagittal imbalance (PI-LL >20° , SVA > 4cm or PT > 20°). Patients were excluded if they had concurrent neurological disorders, other spinal pathologies, or lower limb conditions that could influence gait mechanics. Additionally, individuals with a history of spinal or lower limb surgery were also excluded to minimize confounding factors.
  Interventions: Other: Gait analysis and surface electromyography analysis
- lumbar spinal stenosis Group: This group comprised elderly patients (≥60 years old) clinically diagnosed with lumbar spinal stenosis (LSS) through radiographic findings and symptomatology. Exclusion criteria encompassed: (1) concurrent neurological disorders (e.g., peripheral neuropathy, cerebrovascular disease); (2) comorbid spinal pathologies (e.g., degenerative scoliosis, spondylolisthesis); (3) lower extremity conditions potentially impacting gait biomechanics (e.g., severe osteoarthritis, prior arthroplasty); and (4) any history of spinal or lower limb surgical interventions, thereby minimizing potential confounders.
  Interventions: Other: Gait analysis and surface electromyography analysis
- Lumbar disc herniation Group: This group comprised elderly patients (≥60 years old) clinically diagnosed with Lumbar disc herniation (LDH) through radiographic findings and symptomatology. Exclusion criteria encompassed: (1) concurrent neurological disorders (e.g., peripheral neuropathy, cerebrovascular disease); (2) comorbid spinal pathologies (e.g., degenerative scoliosis, spondylolisthesis); (3) lower extremity conditions potentially impacting gait biomechanics (e.g., severe osteoarthritis, prior arthroplasty); and (4) any history of spinal or lower limb surgical interventions, thereby minimizing potential confounders.
  Interventions: Other: Gait analysis and surface electromyography analysis
- Cervical Spondylosis with Myelopathy Group: This group comprised elderly patients (≥60 years old) clinically diagnosed with Cervical Spondylosis with Myelopathy Group through radiographic findings and symptomatology. Exclusion criteria encompassed: (1) concurrent neurological disorders (e.g., peripheral neuropathy, cerebrovascular disease); (2) comorbid spinal pathologies (e.g., degenerative scoliosis, spondylolisthesis); (3) lower extremity conditions potentially impacting gait biomechanics (e.g., severe osteoarthritis, prior arthroplasty); and (4) any history of spinal or lower limb surgical interventions, thereby minimizing potential confounders.
  Interventions: Other: Gait analysis and surface electromyography analysis
- Healthy Volunteer Group: This group comprised healthy elderly patients (≥60 years old) . Exclusion criteria encompassed: (1) concurrent neurological disorders (e.g., peripheral neuropathy, cerebrovascular disease); (2) comorbid spinal pathologies (e.g., degenerative scoliosis, LSS, LDH, spondylolisthesis); (3) lower extremity conditions potentially impacting gait biomechanics (e.g., severe osteoarthritis, prior arthroplasty); and (4) any history of spinal or lower limb surgical interventions, thereby minimizing potential confounders.
  Interventions: Other: Gait analysis and surface electromyography analysis

INTERVENTIONS:
Other: Gait analysis and surface electromyography analysis — A comprehensive motion analysis system was employed to assess biomechanical parameters during functional tasks. Ground reaction forces (GRFs) were measured using an instrumented force plate, while muscle activation patterns were recorded via surface electromyography (sEMG). Three-dimensional kinematic data were concurrently captured using motion-capture cameras. The standardized testing protocol consisted of: (1) quiet standing (30-second trial) and (2) three consecutive back-and-forth walking cycles (5-meter walkway), enabling the quantification of both static postural control and dynamic gait characteristics.

SUMMARY:
This cross-sectional observational study aims to quantitatively compare three-dimensional gait parameters, surface electromyography (EMG) patterns, and radiological parameters among patients with different degenerative spinal conditions-including lumbar disc herniation (LDH), lumbar spinal stenosis (LSS), lumbar sagittal imbalance (LSI), degenerative lumbar scoliosis (DLS), and cervical spondylotic myelopathy (CSM)-alongside a healthy control group. The analysis focuses on spatiotemporal gait characteristics (step length, stride length, cadence), lower limb kinematics and kinetics (hip/knee/ankle joint angles, moments, and powers during stance and swing phases), and surface EMG amplitudes (thoracic erector spinae, multifidus, gluteus maximus, and rectus abdominis muscles) during standardized walking tasks. Additionally, radiological parameters (e.g., pelvic incidence-lumbar lordosis mismatch, C2-C7 sagittal vertical axis, coronal Cobb angle) will be correlated with gait and muscle activation deviations. The study employs motion capture systems, force plates, and high-density EMG to objectively differentiate disease-specific movement impairments. Findings from this study may establish biomechanical and neuromuscular signatures for each degenerative condition, providing a framework for personalized rehabilitation strategies, gait retraining, and surgical outcome assessment in spinal disorders. Comparative analysis with healthy controls will further elucidate pathological alterations in gait and muscle recruitment patterns caused by degenerative spinal diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the following single disease: degenerative scoliosis, coronal imbalance, lumbar spinal stenosis, lumbar disc herniation, spinal cord-type cervical spondylosis;
2. Age ≥ 60 years, regardless of gender;
3. Planned to undergo elective open spinal fusion surgery;
4. Voluntarily participate in the study, understand and agree to the study content, and sign the informed consent form.

Exclusion Criteria:

1. History of previous spinal surgery;
2. Combined with other neuromuscular diseases (such as Parkinson's disease), inflammatory diseases (such as ankylosing spondylitis), infectious diseases (such as spinal tuberculosis), sepsis, tumors, or lower limb joint diseases that may cause low back and lower limb pain, affecting physical activity;
3. Suffering from severe cardiovascular, cerebral, liver, or kidney disease;
4. Suffering from mental illness, dementia, or unable to cooperate to complete clinical research.

   * Skin rupture in the waist;

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included patients who required surgical treatment at the Spine Research Center for the Elderly at Xuanwu Hospital, Capital Medical University in Beijing, China, as well as healthy volunteers collected in the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Velocity | one week before surgery
  velocity refers to the distance traveled by the human body per unit time during walking and is one of the core parameters for evaluating dynamic gait characteristics.
Cadence | one week before surgery
  Cadence is one of the core spatiotemporal parameters in three-dimensional gait analysis, referring to the number of steps per minute (Steps Per Minute, SPM), which reflects walking rhythm and movement efficiency.
Stride time | one week before surgery
  In three-dimensional gait analysis, stride time refers to the time interval between two consecutive initial contacts of the same heel, representing the duration required to complete a full stride (unit: seconds). Its calculation encompasses both the stance phase and swing phase of a single lower limb, making it one of the core temporal parameters of the gait cycle.
Stance time | one week before surgery
  Stance Time is one of the key spatiotemporal parameters in gait analysis, referring to the period from the initial contact of a single foot with the ground to its complete toe-off. It reflects the weight-bearing and stability performance of the lower limb during the walking cycle.
Swing time | one week before surgery
  The swing phase is a stage in the gait cycle, referring to the time interval from when the foot leaves the ground (toe-off) to when the same foot touches the ground again (heel strike).
Stance phase | one week before surgery
  The Stance Phase refers to the entire stage in the Gait Cycle when the foot is in contact with the ground, starting from Initial Contact (heel strike) and ending with Toe-Off (toe lift) of the same foot. It accounts for approximately 60%~65% of a normal gait cycle (reduced to about 40% during running).
Swing phase | one week before surgery
  Swing Phase is a critical stage in the Gait Cycle, referring to the movement process from when the foot leaves the ground and swings forward until it makes contact with the ground again. During this phase, the lower limb completes actions such as acceleration and deceleration in the air, as well as preparing for the next support phase. In three-dimensional gait analysis, the Swing Phase is quantified using motion capture systems (such as marker points, force plates, and surface electromyography) to measure joint angles, muscle activity, and spatiotemporal parameters, providing objective data for clinical gait assessment.
Single support phase | one week before surgery
  Single Support Phase is a critical stage in the Gait Cycle, referring to the period when one foot fully bears the body weight while the other lower limb is in the Swing Phase.
Double support phase | one week before surgery
  The Double Support Phase is a crucial time stage in the gait cycle, referring to the moment during walking when both feet are simultaneously in contact with the ground. This phase holds significant importance in gait analysis, particularly in 3D Gait Analysis, where it is used to assess balance, gait stability, and neuromuscular control.
Stride length | one week before surgery
  Stride Length refers to the horizontal distance between two consecutive points of contact by the same foot. It is a crucial parameter in gait analysis for evaluating the walking cycle, particularly significant in clinical rehabilitation, sports medicine, and biomechanics research.
Step length | one week before surgery
  Step length refers to the horizontal distance between two consecutive ground contact points of the heel on the same side (i.e., the forward distance from the previous heel contact point to the next heel contact point when the left/right foot takes a step).
Step Width | one week before surgery
  Step Width is a crucial parameter in Gait Analysis, used to quantify gait stability and balance control during human walking. It holds significant clinical value, particularly in fields such as neuromuscular disorders, fall risk assessment, and sports injury rehabilitation.
Gait Deviation Index | one week before surgery
  The Gait Deviation Index is a standardized metric used to quantitatively assess the degree of gait abnormalities, calculated based on data from 3D motion analysis systems. It is widely applied in rehabilitation medicine, orthopedics, and neuroscience, particularly for gait analysis in patients with conditions such as cerebral palsy, stroke, and spinal cord injuries.
Hip Range of Motion | one week before surgery
  Hip joint range of motion refers to the dynamic angular changes of the hip joint in three planes of movement, quantitatively measured using a motion capture system during three-dimensional gait analysis (3D Gait Analysis). It is a critical parameter for assessing gait abnormalities, hip joint function, and neuromuscular disorders.
Knee Range of Motion | one week before surgery
  Knee range of motion refers to the dynamic movement range of the knee joint in the sagittal, coronal, and transverse planes quantitatively measured by a motion capture system during three-dimensional gait analysis. It is one of the core parameters for evaluating walking function, joint stability, and postoperative rehabilitation outcomes.
Ankle Range of Motion | one week before surgery
  Ankle range of motion (AROM) refers to the dynamic movement range of the ankle joint during the gait cycle, typically quantified and assessed in three dimensions: the sagittal plane (flexion-extension), the coronal plane (inversion-eversion), and the horizontal plane (internal-external rotation). It holds significant importance for diagnosing gait abnormalities, monitoring rehabilitation outcomes, and surgical planning.
Hip joint moment | one week before surgery
  Hip joint moment refers to the biomechanical load acting on the hip joint during the gait cycle, reflecting the mechanical balance of muscles, ligaments, and bones around the joint. In three-dimensional gait analysis, it is calculated using dynamic models, with units in newton-meters (N·m) or normalized to body weight multiples (N·m/kg).
Knee joint moment | one week before surgery
  Knee joint moment is a key dynamic parameter in gait analysis, referring to the rotational force (torque) acting on the knee joint during walking or movement, which reflects the mechanical load state of the muscles, ligaments, and bones around the knee joint.
Ankle joint moment | one week before surgery
  Ankle Joint Moment refers to the internal and external moments acting on the ankle joint in the sagittal, coronal, and horizontal planes, calculated through combined measurements using a 3D motion capture system and force plates during gait analysis. It reflects the dynamic load state of the muscles, ligaments, and skeletal structures surrounding the ankle joint.
Average EMG | one week before surgery
  Average EMG (AEMG) refers to the average amplitude value of the electrical signals from the target muscle collected via surface electromyography (sEMG) after rectification and filtering during a gait cycle (or a specific time period) in three-dimensional gait analysis, reflecting the overall intensity of muscle activity.
Integrated electromyography | one week before surgery
  The integrated electromyography (iEMG) is a quantitative metric in surface electromyography (sEMG) analysis, referring to the cumulative sum of EMG signal amplitudes over a specific time period, reflecting the overall intensity of muscle activity. In three-dimensional gait analysis, iEMG is commonly used to assess the synergistic activation patterns and fatigue levels of different muscles during the walking cycle.
Root mean square | one week before surgery
  The root mean square (RMS) average of surface electromyography is a time-domain analysis method used in surface electromyography (sEMG) signal processing to quantify the electrical activity intensity of muscles during specific movements (such as walking or running).
The maximum root mean square of surface electromyography | one week before surgery
  The maximum root mean square of surface electromyography (RMSmax) refers to the maximum activation intensity value (unit: μV or mV) of a specific muscle during the gait cycle, obtained by processing the muscle's electrical signals collected via surface electrodes using root mean square (RMS) analysis in three-dimensional gait analysis.
Mean Power Frequency | one week before surgery
  Mean Power Frequency (MPF) is one of the key indicators in the frequency domain analysis of surface electromyography (sEMG), reflecting the main frequency energy distribution of motor unit action potentials (MUAPs) during muscle contraction. In 3D gait analysis, MPF is used to quantify muscle fatigue levels, neuromuscular control strategies, and functional movement states.
Median Frequency | one week before surgery
  The median frequency of surface electromyography (sEMG) refers to the frequency point in the power spectrum where the total energy is divided into two equal parts (i.e., 50% of the energy lies above and below this frequency) through spectral analysis of the EMG signal (typically using Fast Fourier Transform, FFT).

SECONDARY OUTCOMES:
Visual Analogue Scale | one week before surgery
  VAS assessment uses a straight line or ruler about 10 centimeters long, with one end marked as 0 and the other as 10. 0 represents no pain, and 10 represents the most severe pain. The patient marks a point on the line according to their pain perception, and this point represents the patient's pain intensity.
Oswestry disability index | one week before surgery
  The validated ODI is a self-administered questionnaire for evaluating back-specific functional disability, consisting of 10 items with scores from 0 to 5, and higher ODI indicates more severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No